CLINICAL TRIAL: NCT07024095
Title: "Effects of Inspiratory Muscle Training on Pulmonary Function, Functional Capacity, and Quality of Life After Percutaneous Vertebroplasty in Individuals With Osteoporotic Vertebral Compression Fracture"
Brief Title: Inspiratory Muscle Training After Vertebroplasty in Osteoporotic Fracture Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISTÜ-IMT-001
Record Dates: First submitted 2025-06-03; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Osteoporotic Vertebral Compression Fractures; Restrictive Pulmonary Disorders; Inspiratory Muscle Weakness; Postoperative Pulmonary Function
Keywords: Vertebroplasty; Functional Capacity; Respiratory Muscle Training; Rehabilitation; Physical Fitness
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two parallel groups using stratified randomization based on potential confounding variables such as age and sex:
  * The intervention group will receive inspiratory muscle training (IMT) in addition to standard postoperative rehabilitation.
  * The control group will receive only standard postoperative rehabilitation.
  Randomization will be performed using a computer-generated stratified sequence, and group allocation will be concealed. The interventions will be conducted in parallel over a period of 8 weeks.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded to their group assignment to reduce bias related to perception and response. Outcome assessors will also be blinded to ensure objective evaluation of study endpoints. Due to the nature of the intervention, care providers and investigators will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İnspiratory traning group (Experimental): Participants in the intervention group will receive, in addition to the standard postoperative follow-up for 8 weeks (3 days per week), a home-based exercise program including diaphragmatic breathing exercises, stretching exercises targeting kyphotic posture, and strengthening exercises for the thoracic region. These exercises will be taught to the patients and their caregivers by a licensed physiotherapist before hospital discharge.
  In addition, inspiratory muscle training (IMT) will be performed every day for 8 weeks. To ensure progressive workload, maximal inspiratory pressure (MIP) will be reassessed weekly, and the IMT device will be adjusted accordingly.
  Interventions: Behavioral: Inspiratory Muscle Training (IMT)
- Control Group (Active Comparator): Participants in the control group will receive, similar to the intervention group, a home-based exercise program for 8 weeks (3 days per week), including diaphragmatic breathing exercises, stretching exercises for kyphotic posture, and strengthening exercises for the thoracic region, in addition to standard postoperative follow-up. These exercises will be demonstrated to the patients and their caregivers by a licensed physiotherapist before hospital discharge.
  Unlike the intervention group, participants in this group will not receive inspiratory muscle training (IMT).
  Interventions: Behavioral: control group

INTERVENTIONS:
Behavioral: Inspiratory Muscle Training (IMT) — Participants in the intervention group will receive, in addition to the standard postoperative follow-up for 8 weeks (3 days per week), a home-based exercise program including diaphragmatic breathing exercises, stretching exercises targeting kyphotic posture, and strengthening exercises for the thoracic region. These exercises will be taught to the patients and their caregivers by a licensed physiotherapist before hospital discharge.
  In addition, inspiratory muscle training (IMT) will be performed every day for 8 weeks. To ensure progressive workload, maximal inspiratory pressure (MIP) will be reassessed weekly, and the IMT device will be adjusted accordingly.
  Arms: İnspiratory traning group
Behavioral: control group — Participants in the control group will receive, similar to the intervention group, a home-based exercise program for 8 weeks (3 days per week), including diaphragmatic breathing exercises, stretching exercises for kyphotic posture, and strengthening exercises for the thoracic region, in addition to standard postoperative follow-up. These exercises will be demonstrated to the patients and their caregivers by a licensed physiotherapist before hospital discharge.
  Unlike the intervention group, participants in this group will not receive inspiratory muscle training (IMT).
  Arms: Control Group

SUMMARY:
This study investigates the long-term effects of inspiratory muscle training (IMT) on pulmonary function, functional capacity, and quality of life in individuals with osteoporotic vertebral compression fractures who have undergone percutaneous vertebroplasty.

Participants aged 50 and older, diagnosed with osteoporosis and having undergone thoracic vertebroplasty within the past 3 months, will be randomly assigned to either an intervention group (IMT + standard rehabilitation) or a control group (standard rehabilitation only).

The primary outcome measure is spirometry-based pulmonary function. Secondary outcome measures include inspiratory muscle strength, functional walking capacity (6-minute walk test), diaphragmatic structure and elasticity, and quality of life (SGRQ, NHP).

This randomized controlled trial will be conducted at the Cardiopulmonary Rehabilitation Unit of Nuh Naci Yazgan University and aims to provide scientific evidence for integrating IMT into routine post-vertebroplasty rehabilitation protocols.

DETAILED DESCRIPTION:
Vertebral compression fractures (VCFs) are among the most common complications of osteoporosis. In a Germany-based study, the annual incidence of VCFs in individuals aged 50 and above was reported as 307 per 100,000 people. The same study estimated the direct healthcare cost of VCFs to be approximately €6,490 within the first year after the fracture. The risk of VCF increases with age in both sexes, with a 40% rise in postmenopausal women. Although there is no specific epidemiological study on the incidence of VCFs in Turkey, a study conducted in 2025 reported an increased incidence of osteoporotic vertebral fractures due to limited access to healthcare and significantly reduced physical activity during the COVID-19 pandemic. Approximately one-third of osteoporotic VCFs are symptomatic and significantly reduce patients' quality of life. Whether symptomatic or asymptomatic, osteoporotic VCFs can lead to various health issues such as spinal deformities, nerve damage, functional limitations in thoracic and abdominal organs, reduced mobility, impaired pulmonary function, depression, and decreased quality of life. These fractures are also a major cause of acute and chronic back pain and are associated with increased risk of new fractures and mortality.

Percutaneous vertebroplasty (PV) is a minimally invasive procedure commonly used in the treatment of spinal pain caused by osteoporotic fractures, vertebral hemangiomas, and metastatic tumors. First performed by Deramond et al. in 1987 for spinal hemangiomas, PV has since been widely adopted as an effective treatment for osteoporotic and neoplastic vertebral fractures. During the procedure, under fluoroscopic or CT guidance, polymethyl methacrylate (PMMA) cement is injected into the fractured or weakened vertebral body through a specialized needle. Early studies reported significant pain reduction following the procedure with rare complications. Even before being fully supported by high-quality randomized controlled trials, PV was incorporated into clinical practice and became part of standard treatment for osteoporotic vertebral fractures. Cadaveric studies have also shown that vertebral body rigidity and mechanical strength are restored following PMMA injection.

Spinal pathologies such as vertebral fractures and deformities are known to cause restrictive pulmonary dysfunctions. Restrictive lung diseases encompass conditions characterized by reduced lung expansion capacity due to etiologies such as pulmonary fibrosis, neuromuscular diseases, and thoracic deformities. These conditions are associated with decreased total lung capacity (TLC), vital capacity (VC), and functional residual capacity (FRC), leading to impaired alveolar ventilation and increased respiratory muscle workload. Vertebral deformities, in particular, restrict chest wall mobility, preventing optimal function of respiratory muscles and reducing ventilatory capacity. The progressive nature of spinal deformities can reduce diaphragmatic mechanical efficiency and increase the work of breathing. Studies have shown a significant correlation between the degree of vertebral deformity and the degree of pulmonary dysfunction. A 2022 systematic review reported that increased Cobb angle in untreated idiopathic scoliosis is inversely related to forced vital capacity (FVC), VC, and TLC. Similarly, another study on adolescents who underwent thoracoplasty surgery for idiopathic scoliosis showed a significant postoperative decline in respiratory function.

Moreover, changes in respiratory function after PV are not solely due to pain reduction and mechanical improvements, but may also be influenced by physiological effects related to the surgery itself. Local tissue trauma during PV may affect the structural and functional integrity of paraspinal muscles in adjacent vertebral segments. This can result in inflammatory responses, spasms, or inhibition of paraspinal muscles, impairing spinal stability and indirectly limiting chest wall mobility. Additionally, protective breathing patterns due to postoperative pain may lead to dominant apical breathing instead of diaphragmatic breathing, causing inefficient respiratory muscle activity and reduced ventilation efficiency. Considering these physiological impacts, targeted inspiratory muscle training (IMT) in the postoperative period is viewed as a clinically important intervention to prevent or mitigate these adverse outcomes.

Although short-term improvements in pulmonary function following PV have been reported, there is no existing study that compares these improvements with healthy individuals. This creates uncertainty in determining the sufficiency and sustainability of post-PV functional gains relative to the pulmonary performance of the general population. Furthermore, most studies evaluating pulmonary function after PV provide limited long-term follow-up data, making it unclear whether the initial improvements are maintained or whether a decline occurs over time. IMT is thought to have the potential to support and enhance pulmonary function in the long term following PV. Studies have shown that IMT improves respiratory muscle strength, thoracic mobility, and dyspnea symptoms in patients undergoing thoracic surgery, and these effects are sustained in long-term follow-ups. Therefore, implementing IMT in patients after PV is clinically important to preserve the surgical gains, reduce pulmonary complications, and improve quality of life.

IMT is a well-established physiotherapeutic method proven effective following thoracic surgeries. It strengthens the respiratory muscles through resistance-based exercises, improving patients' respiratory capacity and functional recovery. Additionally, studies have shown that IMT can significantly improve balance, quality of life, and dyspnea. For example, a study investigating IMT in individuals with spinal cord injury found that six weeks of IMT significantly improved inspiratory muscle strength, quality of life, and pain compared to the placebo group. In another study by Kocjan et al., diaphragmatic thickness was evaluated via ultrasound following thoracic surgery, and a significant correlation between diaphragmatic thickness and balance levels was reported.

IMT has been shown to improve maximal inspiratory pressure and respiratory muscle endurance, thereby increasing exercise tolerance. Studies in patients with restrictive lung diseases also report that IMT enhances lung compliance and gas exchange efficiency, supporting ventilation-perfusion matching. In a study by Çalık et al., an 8-week IMT program in individuals with ankylosing spondylitis significantly improved respiratory muscle strength, functional exercise capacity, and Ankylosing Spondylitis Disease Activity Index scores. In another study evaluating paraplegic patients using wheelchairs following spinal cord injury, IMT led to significant improvements in aerobic capacity, respiratory muscle strength, and dyspnea compared to the control group.

Although the effects of respiratory muscle training on pulmonary function, muscle strength, quality of life, and balance have been studied in various restrictive pulmonary conditions, no study has evaluated its impact after PV. Therefore, this study aims to investigate the long-term effects of inspiratory muscle training on pulmonary function, inspiratory muscle strength, and quality of life in individuals who have undergone percutaneous vertebroplasty. It is anticipated that IMT may improve respiratory function by reducing dyspnea and enhance quality of life. Additionally, by reducing pulmonary complications, IMT may lead to decreased hospital admissions and lower healthcare costs. Given the limited literature evaluating the effects of IMT after PV, this study may provide a valuable contribution to the scientific literature and support the development of clinical rehabilitation protocols.

ELIGIBILITY:
Inclusion Criteria:

* Being 50 years of age or older at the time of the study,
* Having a diagnosis of osteoporosis confirmed by a specialist physician,
* Having undergone percutaneous vertebroplasty surgery due to an osteoporotic vertebral compression fracture in the thoracic region within the past 3 months,
* Being cooperative with the questionnaires and assessment methods to be used in the study,
* Being able to read and voluntarily agree to participate in the study by signing the informed consent form.

Exclusion Criteria:

* Having a history of diagnosed unstable cardiac disease,
* Having a diagnosed pulmonary or neurological disorder,
* Having experienced an acute infection within the past 15 days,
* Being unable to participate in exercise interventions due to mental or cognitive impairment.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of Forced Vital Capacity - FVC | Baseline, Week 4, and Week 8
  Forced vital capacity (FVC) will be assessed using a Cosmed Pony FX spirometer (Rome, Italy). All measurements will be conducted in accordance with the standards of the European Respiratory Society (ERS) and American Thoracic Society (ATS), with participants seated during the procedure. Each participant will perform at least three acceptable maneuvers, and the highest value will be recorded for analysis. FVC results will be expressed both in liters (L) as absolute values and as percentage of predicted values based on reference equations (Miller et al., 2005). In addition, the lower limit of normal (LLN) for FVC will be calculated (Hankinson et al., 1999).

SECONDARY OUTCOMES:
Assessment Forced Expiratory Volume in 1 Second (FEV1) | Baseline, week 4, week 8
  FEV1 will be measured using the Cosmed Pony FX spirometer following ERS/ATS standardized procedures. Participants will be instructed to perform at least three acceptable maneuvers, and the highest FEV1 value will be used for analysis. Results will be presented as liters (L) and as percent of predicted values based on standardized reference equations. The lower limit of normal (LLN) for FEV1 will also be determined (Hankinson et al., 1999).
Assessment FEV1/FVC Ratio | Baseline, week 4, week 8
  The FEV1/FVC ratio will be calculated using data obtained from spirometric testing with the Cosmed Pony FX spirometer. This parameter will be expressed as a percentage (%), and it will be used to assess the degree of airflow obstruction. Lower values of the FEV1/FVC ratio are indicative of obstructive respiratory patterns.
Assessment Peak Expiratory Flow (PEF) | Baseline, week 4, week 8
  Peak expiratory flow (PEF) will be measured to determine the maximum speed of expiration. Measurements will be conducted using the Cosmed Pony FX spirometer in accordance with ERS/ATS guidelines. PEF values will be expressed in liters per second (L/s). Higher values reflect better expiratory performance.
Assessment of Forced Expiratory Flow at 25-75% of Exhalation (FEF25-75) | Baseline, week 4, week 8
  FEF25-75 will be measured using the Cosmed Pony FX spirometer to assess mid-expiratory flow, which reflects small airway function. Participants will perform multiple spirometric maneuvers, and the highest acceptable value will be used in analysis. Results will be reported in liters per second (L/s).
Assessment of Respiratory Muscle Strength | Baseline, Week 4, and Week 8
  Maximum inspiratory pressure (MIP) and maximum expiratory pressure (MEP) will be measured using an electronic mouth pressure device (Cosmed Pony FX Spirometer, Rome, Italy). MIP and MEP represent intraoral pressures generated against a closed valve and indirectly reflect respiratory muscle strength. For MIP, participants will exhale fully, then perform a maximal inspiratory effort against a closed valve for 1-3 seconds (Graham et al., 2019). For MEP, they will inhale fully and then exhale maximally for about 2 seconds against a closed valve (Miller et al., 2005). At least three acceptable attempts will be recorded for each measure, with a ≤5% difference between the two best values. The highest value will be used for analysis. Age- and sex-based interpretation will be done using reference equations developed by Black and Hyatt (1969).
Assessment of Diaphragm Muscle Thickness | Baseline and Week 8
  To evaluate the morphological characteristics of the diaphragm muscle, high-resolution thoracic computed tomography (CT) images will be used. Images will be acquired using a Siemens CT scanner, and measurements will be taken from the crural region of the diaphragm in axial and coronal planes. Three measurements will be performed for both the right and left hemidiaphragm, and the average values will be recorded. Thickness will be measured from anatomical planes where the muscle borders are clearly defined. Symmetry, atrophy, and positional variations will also be evaluated. All images will be archived in the hospital's PACS system and analyzed by an experienced radiologist using standard anatomical landmarks to ensure reproducibility (Laghi et al., 2021). Diaphragm imaging will be performed during clinically indicated thoracic CT scans conducted as part of routine follow-up after percutaneous vertebroplasty. No additional imaging will be performed for research purposes.
Assessment of Diaphragm Muscle Elasticity | Baseline and Week 8
  To assess the elastic properties of the diaphragm muscle, two-dimensional shear wave elastography (2D-SWE) will be used. Measurements will be performed using a Supersonic Imagine ultrasound device (Aixplorer, Provence, France) equipped with a high-frequency (4-15 MHz) linear probe. Participants will be positioned in the left lateral decubitus position, and the probe will be placed between the 6th and 12th intercostal spaces along the anterior to mid-axillary line to optimally visualize the right hemidiaphragm dome. Once an appropriate image is obtained, the elastography mode will be activated and the elasticity scale set to 0-160 kPa. Participants will be asked to hold their breath at the end of a calm full inspiration. Using the Q-BOX tool, three measurements of diaphragm stiffness will be taken within a 1 mm circular region of interest (ROI), and the mean value will be recorded (Chen et al., 2022).
Assessment of Functional Capacity | Baseline, Week 4, and Week 8
  Functional capacity will be evaluated using the 6-Minute Walk Test (6MWT). Participants will be instructed to walk along a 30-meter flat corridor at the fastest pace they can maintain without running. Standardized verbal encouragement will be provided throughout the test to maintain participant motivation.
  The assessment will be performed twice with a 30-minute interval, and the total distance covered during the second test will be recorded in meters (Enright, 2003). In addition, heart rate, blood pressure, respiratory rate, and oxygen saturation (measured using the Cosmed Spiropalm 6MWT, Rome, Italy) will be recorded before and after the test. Perceived dyspnea and fatigue levels during exertion will be assessed using the Modified Borg Scale (Borg, 1982).
Assessment of Quality of Life | Baseline, Week 4, and Week 8
  Health-related quality of life of the individuals will be assessed using the St. George's Respiratory Questionnaire (SGRQ). This questionnaire consists of 76 items divided into three subscales: Symptoms (29 items), Activity (9 items), and Impacts (38 items). The Symptoms subscale evaluates respiratory complaints such as sputum production, coughing, and shortness of breath. The Activity subscale assesses limitations experienced during physical activities due to breathlessness, while the Impacts subscale examines the broader effects of the disease on daily life and psychosocial functioning. Each subscale, as well as the total score, ranges from 0 to 100, where 0 indicates no impairment in quality of life and 100 indicates severe impairment. The Turkish version of the questionnaire, which has been validated and shown to be reliable, will be used in this study.
Assessment of Quality of Life | Baseline, Week 4, and Week 8
  Perceived health status of the individuals will be assessed using the Nottingham Health Profile (NHP). This questionnaire consists of six subscales: pain, emotional reactions, social isolation, sleep, energy level, and physical mobility. Each subscale evaluates the extent to which the individual is affected in that specific domain of health. Scores for each subscale range from 0 to 100, with higher scores indicating greater negative impact on the individual's health status. The validated and reliable Turkish version of the questionnaire will be used in this study.
Assessment of Kinesiophobia | Baseline, Week 4, and Week 8
  Fear of movement due to pain among study participants will be assessed using the Tampa Scale for Kinesiophobia (TSK). The TSK is a self-report questionnaire designed to evaluate individuals' fear and avoidance behaviors related to physical activity.
  The scale consists of 17 items, each rated on a 4-point Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree). Total scores range from 17 to 68, with higher scores indicating greater levels of kinesiophobia.
  In this study, the Turkish version of the TSK, which has been validated for reliability and cultural relevance, will be used (Yılmaz et al., 2011).

CONTACTS AND LOCATIONS:
Locations (1):
- Nuh Naci Yazgan University, Faculty of Health Sciences - Cardiopulmonary Rehabilitation Unit, Kayseri, Kocasinan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhao H, He Y, Yang JS, Bao W, Chen J, Liu JJ, Li QD, Liu P, Qian B, Zhao YT, Hao DJ. Can paraspinal muscle degeneration be a reason for refractures after percutaneous kyphoplasty? A magnetic resonance imaging observation. J Orthop Surg Res. 2021 Aug 3;16(1):476. doi: 10.1186/s13018-021-02623-y. PMID 34344407
- [Background] Wang B, Zhao CP, Song LX, Zhu L. Balloon kyphoplasty versus percutaneous vertebroplasty for osteoporotic vertebral compression fracture: a meta-analysis and systematic review. J Orthop Surg Res. 2018 Oct 22;13(1):264. doi: 10.1186/s13018-018-0952-5. PMID 30348192
- [Background] Vasold KL, Parks AC, Phelan DML, Pontifex MB, Pivarnik JM. Reliability and Validity of Commercially Available Low-Cost Bioelectrical Impedance Analysis. Int J Sport Nutr Exerc Metab. 2019 Jul 1;29(4):406-410. doi: 10.1123/ijsnem.2018-0283. PMID 30507268
- [Background] Tomas-Carus P, Biehl-Printes C, Del Pozo-Cruz J, Parraca JA, Folgado H, Perez-Sousa MA. Effects of respiratory muscle training on respiratory efficiency and health-related quality of life in sedentary women with fibromyalgia: a randomised controlled trial. Clin Exp Rheumatol. 2022 Jun;40(6):1119-1126. doi: 10.55563/clinexprheumatol/0v55nh. Epub 2022 Jun 22. PMID 35748715
- [Background] Soumyashree S, Kaur J. Effect of inspiratory muscle training (IMT) on aerobic capacity, respiratory muscle strength and rate of perceived exertion in paraplegics. J Spinal Cord Med. 2020 Jan;43(1):53-59. doi: 10.1080/10790268.2018.1462618. Epub 2018 Apr 18. PMID 29667507
- [Background] Robinson HC. Respiratory Conditions Update: Restrictive Lung Disease. FP Essent. 2016 Sep;448:29-34. PMID 27576233
- [Background] Polatli M, Yorgancioglu A, Aydemir O, Yilmaz Demirci N, Kirkil G, Atis Nayci S, Kokturk N, Uysal A, Akdemir SE, Ozgur ES, Gunakan G. [Validity and reliability of Turkish version of St. George's respiratory questionnaire]. Tuberk Toraks. 2013;61(2):81-7. doi: 10.5578/tt.5404. Turkish. PMID 23875584
- [Background] Pazzianotto-Forti EM, da Costa Munno CM, Merino DFB, Simoes da Rocha MR, de Mori TA, Junior IR. Effects of Inspiratory Exercise With Linear and Nonlinear Load on Respiratory Variables Post-Bariatric Surgery. Respir Care. 2019 Dec;64(12):1516-1522. doi: 10.4187/respcare.05841. Epub 2019 Aug 6. PMID 31387894
- [Background] Palermo AE, Cahalin LP, Nash MS. A case for inspiratory muscle training in SCI: potential role as a preventative tool in infectious respiratory diseases like COVID-19. Spinal Cord Ser Cases. 2020 Sep 17;6(1):87. doi: 10.1038/s41394-020-00337-7. PMID 32943611
- [Background] Noonan AM, Brown SHM. Paraspinal muscle pathophysiology associated with low back pain and spine degenerative disorders. JOR Spine. 2021 Sep 15;4(3):e1171. doi: 10.1002/jsp2.1171. eCollection 2021 Sep. PMID 34611593
- [Background] Newall C, Stockley RA, Hill SL. Exercise training and inspiratory muscle training in patients with bronchiectasis. Thorax. 2005 Nov;60(11):943-8. doi: 10.1136/thx.2004.028928. Epub 2005 Jun 30. PMID 15994254
- [Background] Mills DE, Johnson MA, Barnett YA, Smith WH, Sharpe GR. The effects of inspiratory muscle training in older adults. Med Sci Sports Exerc. 2015 Apr;47(4):691-7. doi: 10.1249/MSS.0000000000000474. PMID 25116085
- [Background] Miller MR, Crapo R, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. General considerations for lung function testing. Eur Respir J. 2005 Jul;26(1):153-61. doi: 10.1183/09031936.05.00034505. No abstract available. PMID 15994402
- [Background] Messaggi-Sartor M, Marco E, Martinez-Tellez E, Rodriguez-Fuster A, Palomares C, Chiarella S, Muniesa JM, Orozco-Levi M, Barreiro E, Guell MR. Combined aerobic exercise and high-intensity respiratory muscle training in patients surgically treated for non-small cell lung cancer: a pilot randomized clinical trial. Eur J Phys Rehabil Med. 2019 Feb;55(1):113-122. doi: 10.23736/S1973-9087.18.05156-0. Epub 2018 Jul 6. PMID 29984565
- [Background] Liu JF, Kuo NY, Fang TP, Chen JO, Lu HI, Lin HL. A six-week inspiratory muscle training and aerobic exercise improves respiratory muscle strength and exercise capacity in lung cancer patients after video-assisted thoracoscopic surgery: A randomized controlled trial. Clin Rehabil. 2021 Jun;35(6):840-850. doi: 10.1177/0269215520980138. Epub 2020 Dec 14. PMID 33307766
- [Background] Leake CB, Brinjikji W, Cloft HJ, Kallmes DF. Trends of inpatient spine augmentation: 2001-2008. AJNR Am J Neuroradiol. 2011 Sep;32(8):1464-8. doi: 10.3174/ajnr.A2503. Epub 2011 May 26. PMID 21622578
- [Background] Le Corroller T, Arrigoni F. ESR Essentials: percutaneous bone consolidation-practice recommendations by the European Society of Musculoskeletal Radiology. Eur Radiol. 2025 Sep;35(9):5369-5380. doi: 10.1007/s00330-025-11478-4. Epub 2025 Mar 6. PMID 40050453
- [Background] Lau E, Ong K, Kurtz S, Schmier J, Edidin A. Mortality following the diagnosis of a vertebral compression fracture in the Medicare population. J Bone Joint Surg Am. 2008 Jul;90(7):1479-86. doi: 10.2106/JBJS.G.00675. PMID 18594096
- [Background] Lane JM, Nydick M. Osteoporosis: current modes of prevention and treatment. J Am Acad Orthop Surg. 1999 Jan;7(1):19-31. doi: 10.5435/00124635-199901000-00003. PMID 9916187
- [Background] Laghi FA Jr, Saad M, Shaikh H. Ultrasound and non-ultrasound imaging techniques in the assessment of diaphragmatic dysfunction. BMC Pulm Med. 2021 Mar 15;21(1):85. doi: 10.1186/s12890-021-01441-6. PMID 33722215
- [Background] Kucukdeveci AA, McKenna SP, Kutlay S, Gursel Y, Whalley D, Arasil T. The development and psychometric assessment of the Turkish version of the Nottingham Health Profile. Int J Rehabil Res. 2000 Mar;23(1):31-8. doi: 10.1097/00004356-200023010-00004. PMID 10826123
- [Background] Kumar V, Vatkar AJ, Baburaj V, Najjar E, Bansal P. Pulmonary function after thoracoplasty for adolescent idiopathic scoliosis: a systematic review and meta-analysis. Eur Spine J. 2022 Nov;31(11):2972-2986. doi: 10.1007/s00586-022-07375-9. Epub 2022 Sep 7. PMID 36069937
- [Background] Kumar K, Verma AK, Wilson J, LaFontaine A. Vertebroplasty in osteoporotic spine fractures: a quality of life assessment. Can J Neurol Sci. 2005 Nov;32(4):487-95. doi: 10.1017/s0317167100004492. PMID 16408580
- [Background] Kocjan J, Gzik-Zroska B, Nowakowska K, Burkacki M, Suchon S, Michnik R, Czyzewski D, Adamek M. Impact of diaphragm function parameters on balance maintenance. PLoS One. 2018 Dec 28;13(12):e0208697. doi: 10.1371/journal.pone.0208697. eCollection 2018. PMID 30592726
- [Background] Kempen DHR, Heemskerk JL, Kacmaz G, Altena MC, Reesink HJ, Vanhommerig JW, Willigenburg NW. Pulmonary function in children and adolescents with untreated idiopathic scoliosis: a systematic review with meta-regression analysis. Spine J. 2022 Jul;22(7):1178-1190. doi: 10.1016/j.spinee.2021.12.011. Epub 2021 Dec 25. PMID 34963629
- [Background] Kanis JA. Assessment of fracture risk and its application to screening for postmenopausal osteoporosis: synopsis of a WHO report. WHO Study Group. Osteoporos Int. 1994 Nov;4(6):368-81. doi: 10.1007/BF01622200. PMID 7696835
- [Background] Jung JH, Kim NS. Changes in training posture induce changes in the chest wall movement and respiratory muscle activation during respiratory muscle training. J Exerc Rehabil. 2018 Oct 31;14(5):771-777. doi: 10.12965/jer.1836366.183. eCollection 2018 Oct. PMID 30443522
- [Background] Jones PW, Quirk FH, Baveystock CM, Littlejohns P. A self-complete measure of health status for chronic airflow limitation. The St. George's Respiratory Questionnaire. Am Rev Respir Dis. 1992 Jun;145(6):1321-7. doi: 10.1164/ajrccm/145.6.1321. PMID 1595997
- [Background] Hernlund E, Svedbom A, Ivergard M, Compston J, Cooper C, Stenmark J, McCloskey EV, Jonsson B, Kanis JA. Osteoporosis in the European Union: medical management, epidemiology and economic burden. A report prepared in collaboration with the International Osteoporosis Foundation (IOF) and the European Federation of Pharmaceutical Industry Associations (EFPIA). Arch Osteoporos. 2013;8(1):136. doi: 10.1007/s11657-013-0136-1. Epub 2013 Oct 11. PMID 24113837
- [Background] Hankinson JL, Odencrantz JR, Fedan KB. Spirometric reference values from a sample of the general U.S. population. Am J Respir Crit Care Med. 1999 Jan;159(1):179-87. doi: 10.1164/ajrccm.159.1.9712108. PMID 9872837
- [Background] Graham BL, Steenbruggen I, Miller MR, Barjaktarevic IZ, Cooper BG, Hall GL, Hallstrand TS, Kaminsky DA, McCarthy K, McCormack MC, Oropez CE, Rosenfeld M, Stanojevic S, Swanney MP, Thompson BR. Standardization of Spirometry 2019 Update. An Official American Thoracic Society and European Respiratory Society Technical Statement. Am J Respir Crit Care Med. 2019 Oct 15;200(8):e70-e88. doi: 10.1164/rccm.201908-1590ST. PMID 31613151
- [Background] Galibert P, Deramond H, Rosat P, Le Gars D. [Preliminary note on the treatment of vertebral angioma by percutaneous acrylic vertebroplasty]. Neurochirurgie. 1987;33(2):166-8. French. PMID 3600949
- [Background] Flegal KM. Body-mass index and all-cause mortality. Lancet. 2017 Jun 10;389(10086):2284-2285. doi: 10.1016/S0140-6736(17)31437-X. No abstract available. PMID 28612744
- [Background] Enright PL. The six-minute walk test. Respir Care. 2003 Aug;48(8):783-5. PMID 12890299
- [Background] Chen Y, Li J, Dong B, Zhu Z, Lyu G. Two-dimensional shear wave elastography: a new tool for evaluating respiratory muscle stiffness in chronic obstructive pulmonary disease patients. BMC Pulm Med. 2022 Nov 24;22(1):441. doi: 10.1186/s12890-022-02231-4. PMID 36424581
- [Background] Bronheim R, Khan S, Carter E, Sandhaus RA, Raggio C. Scoliosis and Cardiopulmonary Outcomes in Osteogenesis Imperfecta Patients. Spine (Phila Pa 1976). 2019 Aug 1;44(15):1057-1063. doi: 10.1097/BRS.0000000000003012. PMID 31335789
- [Background] Boswell-Ruys CL, Lewis CRH, Wijeysuriya NS, McBain RA, Lee BB, McKenzie DK, Gandevia SC, Butler JE. Impact of respiratory muscle training on respiratory muscle strength, respiratory function and quality of life in individuals with tetraplegia: a randomised clinical trial. Thorax. 2020 Mar;75(3):279-288. doi: 10.1136/thoraxjnl-2019-213917. Epub 2020 Jan 14. PMID 31937553
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Black LF, Hyatt RE. Maximal respiratory pressures: normal values and relationship to age and sex. Am Rev Respir Dis. 1969 May;99(5):696-702. doi: 10.1164/arrd.1969.99.5.696. No abstract available. PMID 5772056
- [Background] Belkoff SM, Mathis JM, Jasper LE, Deramond H. The biomechanics of vertebroplasty. The effect of cement volume on mechanical behavior. Spine (Phila Pa 1976). 2001 Jul 15;26(14):1537-41. doi: 10.1097/00007632-200107150-00007. PMID 11462082
- [Background] Basha MA, Azab AR, Elnaggar RK, Aboelnour NH, Kamel NM, Aloraini SM, Kamel FH. Inspiratory muscle training impact on respiratory muscle strength, pulmonary function, and quality of life in children with chest burn: A randomized controlled trial. Burns. 2024 Sep;50(7):1916-1924. doi: 10.1016/j.burns.2024.05.007. Epub 2024 May 10. PMID 38782684
- [Background] Basbug G, Gurses HN, Zeren M, Elmadag NM. Effects of inspiratory muscle training on respiratory muscle strength, respiratory function and functional capacity in adolescents with idiopathic scoliosis : A randomized, controlled trial. Wien Klin Wochenschr. 2023 Jun;135(11-12):282-290. doi: 10.1007/s00508-023-02197-1. Epub 2023 Apr 18. PMID 37071202
- [Background] Aktan R, Tertemiz KC, Yigit S, Ozalevli S, Ozgen Alpaydin A, Ucan ES. Effects of home-based telerehabilitation-assisted inspiratory muscle training in patients with idiopathic pulmonary fibrosis: A randomized controlled trial. Respirology. 2024 Dec;29(12):1077-1084. doi: 10.1111/resp.14810. Epub 2024 Aug 11. PMID 39129185